CLINICAL TRIAL: NCT06027762
Title: Assessment of Vertical Ground Reaction Force Measurement During Walking With Feetme® Insoles in Healthy Adults
Brief Title: Assessment of vGRF Measurement During Walking With Feetme® Insoles in Healthy Adults
Acronym: FeetMe-GRF
Status: Completed | Type: Observational
Sponsor: FeetMe (Industry)
Collaborators: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02409-32
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-Groupe

SUMMARY:
The objective of the present study is to demonstrate the validity and reliability of vGRF and other gait parameters measurement in healthy adults while walking with FeetMe® insoles compared to force plates (AMTI BP400600) and video motion capture system (Vicon NEXUS and MX-T40) .

ELIGIBILITY:
Inclusion Criteria.

Volunteers with following criteria satisfied:

* Between the ages of 18 and 80.
* Shoe size between 35 to 46.
* Body weight from 40kg to 120kg.
* Able to walk for 30 mins without assistance.
* Comfortable with using a smartphone.

Non-inclusion Criteria.

A volunteer will not be included if one of the following conditions is met:

* cognitive or behavioral problems limiting communication or participation in the study
* deprivation of liberty by a legal or administrative decision
* adults subject to a legal protection measure or unable to express their consent
* pregnant, parturient and nursing mothers
* people admitted to a health or social establishment for purposes other than research
* Past or planned surgery with the possibility of impacting walking in the past 3 months or which had an impact on walking: orthopedic surgery, trauma to the lower limbs and spine, urological or gynecological surgery, brain and spinal cord surgery .
* Chronic disease affecting walking: Rheumatological, orthopedic, painful, neurological pathology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults between 18 and 85 years old without gait pathologies
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
precision of measurement of 'maximum weight acceptance' and 'push-off' peaks in healthy adults by FeetMe® insoles | between February 2022 and November 2022
  The primary objective of this clinical trial is to quantify precision of measurement of two peaks of vGRF, peaks that correspond to 'maximum weight acceptance' and 'push-off', also called 'heelmax load' and 'toemax load' for healthy adults by FeetMe® insoles compared with Vicon and force plates during a free walk test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Saint-Maurice, Saint-Maurice, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
legal reasons